CLINICAL TRIAL: NCT06982248
Title: Efficacy of Quercetin Loaded on Chitosan Nanoparticles Gel as an Adjunctive to Mechanical Debridement in Treatment of Periodontitis: Randomized Controlled Clinical Trial
Brief Title: The Proposed Study Aims to Investigate the Efficacy of Quercetin as an Adjunctive to Mechanical Debridement in Treatment of Periodontitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: A03030240H
Record Dates: First submitted 2024-12-11; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket | interventions — Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: Group 1: Periodontitis patients treated by NSPT and chitosan nanoparticles gel loaded by quercetin.
  Group 2: Periodontitis patients treated by NSPT and chitosan nanoparticles gel. Group 3: Periodontitis patients treated by NSPT only. Group 4: Periodontally healthy subjects.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1: Periodontitis patients treated by NSPT and chitosan nanoparticles gel loaded by quercetin (Experimental): selected patients receive SRP and chitosan nanoparticles gel loaded by quercetin
  Interventions: Drug: NSP and chitosan nanoparticles gel loaded by quercetin
- Group 2: Periodontitis patients treated by NSPT and chitosan nanoparticles gel. (Experimental): selected patients receive SRP and chitosan nanoparticles gel
  Interventions: Drug: NSP and chitosan nanoparticles gel
- Group 3: Periodontitis patients treated by NSPT only (Active Comparator): NSPT
  Interventions: Procedure: scaling and root planning
- Group 4: Periodontally healthy subjects. (No Intervention): healthy individual act as control group

INTERVENTIONS:
Drug: NSP and chitosan nanoparticles gel loaded by quercetin — NSP and chitosan nanoparticles gel loaded by quercetin
  Arms: Group 1: Periodontitis patients treated by NSPT and chitosan nanoparticles gel loaded by quercetin
Drug: NSP and chitosan nanoparticles gel — NSP and chitosan nanoparticles gel
  Arms: Group 2: Periodontitis patients treated by NSPT and chitosan nanoparticles gel.
Procedure: scaling and root planning — NSPT
  Arms: Group 3: Periodontitis patients treated by NSPT only

SUMMARY:
the proposed study aims to investigate the effect of Quercetin in treatment of periodontitis patients

DETAILED DESCRIPTION:
the proposed study aims to investigate the effect of Quercetin in treatment of periodontitis patients not having systemic diseases.the 2ry aim of study to estimate the neacular factor kabba B level in gingival crevicular fluids.

ELIGIBILITY:
Inclusion Criteria:

- Patients of both sexes with an age ranging between 25 and 55 years will be included in the study. Patients diagnosed as having periodontitis based on clinical and radiographic examinations will be included

Exclusion Criteria:

* Insulin dependent diabetes
* Thyroid disease
* Patients with sensitivity to the medication used in the study
* patients with a history of antibiotic use or anti-inflammatory drugs during the previous 3 months prior to the study will be excluded from the study.
* Additionally, patients with systemic diseases, smokers, pregnant and lactating patients, and patients not compliant with oral hygiene procedures will also be excluded

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
assessment clinical attachment level by UNC 15 periodontal probe | 12 weeks

SECONDARY OUTCOMES:
assessment of the gingival crevicular levels of NF-κB by Elisa kit | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jilan mohamed, Study Director — Mansoura University
Locations (1):
- Faculty of Dentistry, Mansoura University, Aga, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Clinical effect of Quercetin in treatment of periodiontal pocket